CLINICAL TRIAL: NCT03043599
Title: Consolidative Ipilimumab and Nivolumab With Thoracic Radiotherapy After Platinum Based Chemotherapy for Patients With Extensive-Stage Small Cell Lung Cancer
Brief Title: Ipilimumab + Nivolumab w/Thoracic Radiotherapy for Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18914; CA209-840 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Small Cell Lung Cancer; Extensive-stage Small Cell Lung Cancer
Keywords: Thoracic; Radiotherapy; Platinum Based Chemotherapy; Immunotherapy; Ipilimumab; Nivolumab; Extensive-Stage Disease Small Cell Lung Cancer (ED-SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Radiotherapy; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination Therapy (Experimental): Consolidative Ipilimumab and Nivolumab with Thoracic Radiotherapy after Platinum Based Chemotherapy. Radiotherapy, followed by a 14 to 21 day break between radiotherapy and the beginning of study drug treatment.
  Interventions: Radiation: Thoracic Radiation Therapy; Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Radiation: Thoracic Radiation Therapy — All participants will receive radiation therapy (3Gy x 10 fractions) to the chest for 10 days (Monday through Friday for 2 weeks).
  Other Names: radiotherapy
Drug: Ipilimumab — Ipilimumab 3 mg/kg (90 minute IV infusion) will be administered every 3 weeks for 4 doses.
  Other Names: YERVOY
Drug: Nivolumab — Nivolumab 1 mg/kg (30 minute IV infusion) will be administered every 3 weeks for 4 doses, followed by nivolumab 480 mg every 4 weeks.
  Other Names: OPDIVO

SUMMARY:
The purpose of the safety run in Phase I portion of this study is to confirm the recommended Phase II dose of ipilimumab and nivolumab among participants treated with combined thoracic radiation therapy (30 Gy in 10 fractions) and nivolumab/ipilimumab following standard treatment with 4-6 cycles of platinum-based chemotherapy.

The purpose of the Phase II portion of this study is to estimate the 6-month Progression Free Survival (PFS) rate among participants treated with ipilimumab and nivolumab with thoracic radiation therapy (30 Gy in 10 fractions) after standard treatment with 4 to 6 cycles of platinum based chemotherapy.

DETAILED DESCRIPTION:
This study is a nonrandomized, phase II, single arm, multicenter trial evaluating safety and efficacy of thoracic radiation therapy followed by nivolumab and ipilimumab in participants with Extensive-Stage Disease Small Cell Lung Cancer (ED-SCLC) who have completed a first-line platinum-based chemotherapy regimen and achieved ongoing complete response (CR), partial response (PR), or stable disease (SD). This study will determine whether nivolumab and ipilimumab delivered 2 weeks following consolidative thoracic radiation therapy demonstrates acceptable toxicity and whether the treatment regimen will improve 6-month progression-free survival (PFS) compared with a similar historical control cohort in this participant population. Additional objectives include further characterization of overall survival, adverse event profile, patterns of failure analysis, and potential predictive biomarkers of response to nivolumab in combination with ipilimumab and thoracic radiation therapy in patients with ED-SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
* Patients with Small Cell Lung Cancer (SCLC) documented by histology or cytology from brushing, washing, or needle aspiration of a defined lesion, but not from sputum cytology alone
* Have presented at initial diagnosis with extensive-stage disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Have received 4-6 cycles of platinum-based first-line chemotherapy and have an ongoing response of complete response (CR), partial response (PR), or stable disease (SD) after completion of chemotherapy. Acceptable combinations, as recommended per National Comprehensive Cancer Network (NCCN) guidelines, include cisplatin or carboplatin combined with either etoposide or irinotecan; As an exception to the above criterion, participants receiving only 3 cycles of chemotherapy due to toxicity are eligible, if they have an ongoing PR or CR after the 3rd cycle; Participants who have received > 6 cycles of platinum-based first-line chemotherapy are not eligible.
* Participants must initiate study treatment with thoracic radiation therapy less than or equal to 8 weeks (56 days) from the last dose of platinum-based first line chemotherapy.
* Whenever possible, a formalin-fixed, paraffin-embedded (FFPE) tumor tissue block or 10 unstained slides of tumor sample (archival or recent) for biomarker evaluation should be made available and submitted to the central lab for correlative studies.
* Participant re-enrollment: This study permits the re-enrollment of a participant who has discontinued the study due to pre-treatment failure (i.e., participant has not been treated). If re-enrolled, the participant must be re-consented.
* Men and women at least 18 years of age
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to the start of thoracic radiation therapy
* Women must not be breastfeeding.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 5 half-lives of study drug (half-life up to 25 days) plus 30 days (duration of ovulatory cycle) for a total of 5 months post-treatment completion.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 5 half-lives of the study drug (half-life up to 25 days) plus 90 days (duration of sperm turnover) for a total of 7 months post-treatment completion.
* Additional criteria may apply

Exclusion Criteria:

* Participants with previous brain metastases are eligible provided that they are treated and asymptomatic not requiring steroids or anticonvulsants, and have stable disease at the screening tumor assessment. A 4 week disease stable interval as confirmed by MRI or CT brain with contrast is required after treatment of brain metastases before initiation of thoracic radiation therapy. In addition, participants must have been either off corticosteroids, or on a stable or decreasing dose of 10 mg daily prednisone (or equivalent).
* Participants who have received prior chest radiation which at the discretion of the treating radiation oncologist precludes delivery of protocol radiation therapy
* Carcinomatous meningitis
* Pleural effusion that cannot be controlled with appropriate interventions
* All toxicities attributed to prior anti-cancer therapy must have been resolved to Grade 1 (NCI CTCAE Version 4) or baseline before administration of study drug(s) other than: Patients with toxicities attributed to prior anti-cancer therapy that either are not expected to resolve and/or result in long-lasting sequelae, such as neuropathy after platinum-based therapy, or are not expected to interfere with treatment on study, such as fatigue,alopecia, or grade 2 hematologic toxicity are eligible.
* Women who are pregnant or breastfeeding
* Active, known, or suspected autoimmune disease. Patients with an autoimmune paraneoplastic syndrome requiring concurrent immunosuppressive treatment are excluded. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* A condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Corticosteroids with minimal systemic absorption (inhaled or topical steroids) and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
* Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways)
* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Any patient requiring supplemental oxygen therapy
* Previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period
* Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug(s) administration or interfere with the interpretation of safety results
* Major surgery or significant traumatic injury that is not recovered at least 14 days before the initiation of thoracic radiation therapy.
* Positive test for hepatitis B virus (HBV) using HBV surface antigen (HBVsAg) test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection
* Individuals with a positive test for HCV antibody but no detection of HCV RNA indicating no current infection are eligible
* Known medical history of testing positive for human immunodeficiency virus (HIV) or known medical history of acquired immunodeficiency syndrome (AIDS)
* Inadequate hematologic function according to study guidelines
* Inadequate hepatic function according to study guidelines
* History of allergy or hypersensitivity to any of the study drugs or study drug components
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2023-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradford A. Perez, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Perez BA, Kim S, Wang M, Karimi AM, Powell C, Li J, Dilling TJ, Chiappori A, Latifi K, Rose T, Lannon A, MacMillan G, Saller J, Grass GD, Rosenberg S, Gray J, Haura E, Creelan B, Tanvetyanon T, Saltos A, Shafique M, Boyle TA, Schell MJ, Conejo-Garcia JR, Antonia SJ. Prospective Single-Arm Phase 1 and 2 Study: Ipilimumab and Nivolumab With Thoracic Radiation Therapy After Platinum Chemotherapy in Extensive-Stage Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2021 Feb 1;109(2):425-435. doi: 10.1016/j.ijrobp.2020.09.031. Epub 2020 Sep 28. PMID 33002543

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Therapy
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 11
Age, Continuous [Median (Full Range); unit: years] | 66 [45 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Confirmation of Recommended Phase II Dose
Description: Recommended Phase II dose of ipilimumab and nivolumab among participants treated with combined thoracic radiation therapy (30 Gy in 10 fractions) and nivolumab/ipilimumab following standard treatment with 4-6 cycles of platinum-based chemotherapy. Investigators will initially enroll 6 patients and wait until completion of the 13-week safety observation period following initiation of ipilimumab + nivolumab combination treatment.
Time Frame: 13 weeks
Measure: Number; unit: mg/kg dose
Arm/Group | Combination Therapy
Number analyzed (Participants) | 21
mg/kg dose
  Ipilimumab | 3
  Nivoumab | 1

2. Primary Outcome: Phase II: Progression Free Survival (PFS)
Description: PFS is defined as the duration from date of registration to date of first documentation of progression assessed by local investigator or symptomatic deterioration (as defined above) or death due to any cause.
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 21
months | 4.5 [2.7 to 4.6]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration from date of registration to date of death due to any cause. Participants last known to be alive are censored at date of last contact.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 21
months | 11.7 [4.7 to 16.0]

ADVERSE EVENTS:
Time Frame: 2 years
Description: All Serious Adverse Events are reported, regardless of causality. Serious Adverse Events were reported during screening period and within 100 days of discontinuation of dosing.
Arm/Group | Combination Therapy
All-Cause Mortality (participants affected / at risk) | 6/21
Serious Adverse Events (participants affected / at risk) | 13/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=21)
Diarrhea (Gastrointestinal disorders) | 4 (7)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Neoplasms benign, malignant and unspecified -Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Neck Pain (General disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1) — Urosepsis presumed related to kiebsiella pneumoniae
Lung Infection (Infections and infestations) | 6 (7)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders -Other (Metabolism and nutrition disorders) | 1 (2) — SIADH
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness - lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (3)
Headache (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) — Death due to disease progression
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Death due to lung infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=21)
Hypothyroidism (Endocrine disorders) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 7 (20)
Nausea (Gastrointestinal disorders) | 7 (8)
Fatigue (General disorders) | 6 (8)
Fever (General disorders) | 8 (11)
Weight Loss (Investigations) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
SIADH (Metabolism and nutrition disorders) | 1 (2)
Dizziness (Nervous system disorders) | 7 (8)
Cognitive Disturbance (Nervous system disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Hypertension (Vascular disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 6 (6)
Pain (General disorders) | 5 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 5 (6)
Insomnia (Psychiatric disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 6 (8)
Esophagitis (Gastrointestinal disorders) | 10 (11)
Gait Disturbance (General disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 6 (8)
Headache (Nervous system disorders) | 4 (4)
Confusion (Psychiatric disorders) | 2 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 1 (3)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (5)
Depression (Psychiatric disorders) | 4 (5)
Gynecomastia (Reproductive system and breast disorders) | 1 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Edema Limbs (General disorders) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Infusion related reaction (General disorders) | 1 (1)
Infections and Investigations- Other (Infections and infestations) | 2 (2)
Lung Infection (Infections and infestations) | 6 (9)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (5)
Platelet count decreased (Investigations) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — mouth sores
Memory impairment (Nervous system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Chills (General disorders) | 2 (3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 5 (5)
Bronchial infection (Infections and infestations) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Hypotension (Vascular disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye Disorders - Other (Eye disorders) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash, erythematous (Skin and subcutaneous tissue disorders) | 2 (2)
Metabolism and Nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1) — Alkalosis and hypokalemia attributed to cushings syndrome secondary to ectopic ACTH from SCLC
Neoplasms benign, malignant and unspecified -Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03043599/Prot_SAP_000.pdf